CLINICAL TRIAL: NCT01995123
Title: Behavioral Activation for Smoking Cessation in Veterans With PTSD
Brief Title: Behavioral Activation for Smoking Cessation in PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHBA-002-12F; NCT01947725 (obsolete NCT alias)
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-03

CONDITIONS: Tobacco Dependence; PTSD
Keywords: Tobacco dependence; PTSD; Behavioral Activation Therapy
MeSH Terms: conditions — Tobacco Use Disorder; Stress Disorders, Post-Traumatic | interventions — Health

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral Activation Therapy (Experimental): Behavioral Activation (BA) Treatment will be delivered in eight, 30 minute individual sessions over an 8-week period. BA treatment will focus on encouraging subjects to participate in activities that they find enjoyable and rewarding. In addition, this arm will receive standard smoking cessation therapy, nicotine patch, and either nicotine gum or nicotine lozenge.
  Interventions: Behavioral: Behavioral Activation Therapy; Behavioral: Standard Smoking Cessation Therapy
- Health and Smoking Education (Active Comparator): Health and Smoking Education (HSE) Treatment will be delivered in eight, 30 minute individual sessions over an 8-week period. HSE treatment will focus on smoking, health, and the impact of smoking on the subject's health. In addition, this arm will receive standard smoking cessation therapy, nicotine patch, and either nicotine gum or nicotine lozenge.
  Interventions: Behavioral: Health and Smoking Education; Behavioral: Standard Smoking Cessation Therapy

INTERVENTIONS:
Behavioral: Behavioral Activation Therapy — Behavioral Activation (BA) Treatment will be delivered in eight, 30 minute individual sessions over an 8-week period. BA treatment will focus on encouraging subjects to participate in activities that they find enjoyable and rewarding.
  Arms: Behavioral Activation Therapy
Behavioral: Health and Smoking Education — Health and Smoking Education (HSE) Treatment will be delivered in eight, 30 minute individual sessions over an 8-week period. HSE treatment will focus on smoking, health, and the impact of smoking on the subject's health.
  Arms: Health and Smoking Education
Behavioral: Standard Smoking Cessation Therapy — Standard smoking cessation therapy will be delivered in eight, 20-minute individual sessions over an 8-week period.

SUMMARY:
The purpose of this study is to examine whether behavioral activation as an adjuvant to standard smoking cessation treatment improves smoking cessation outcomes among veterans with PTSD relative to a comparably intense combination of standard smoking cessation treatment + health and smoking education. It is expected that behavioral activation will produce more successful results than health and smoking education when paired with standard smoking cessation treatment.

DETAILED DESCRIPTION:
The purpose of this study is to examine whether behavioral activation as an adjuvant to standard smoking cessation treatment improves smoking cessation outcomes among veterans with PTSD relative to a comparably intense combination of standard smoking cessation treatment + health and smoking education. It is expected that behavioral activation will produce more successful results than health and smoking education when paired with standard smoking cessation treatment.

After an initial phone screen, in-person screening, and baseline assessment, enrolled participants will be randomized to either behavioral activation therapy and standard smoking cessation treatment (BA+ST) or health and smoking education and standard smoking cessation treatment (HSE+ST). Both groups will meet with a therapist once a week for 8 weeks to receive either BA+ST or HSE+ST. Participants' mood and smoking outcomes will be monitored throughout the 8 weeks of treatment and at 2 follow-up visits and 2 follow-up phone calls.

ELIGIBILITY:
Inclusion Criteria:

* Report smoking an average of 10 or more cigarettes daily for at least six months
* Report a desire to quit smoking
* Meet criteria for current PTSD
* Speak and read English
* Agree to participate in the study
* Be 18 years old
* Be a veteran

Exclusion Criteria:

* Meeting criteria for psychotic or bipolar disorder
* Psychoactive substance abuse or dependence (excluding nicotine dependence) within the past 6 months
* Inability to give informed, voluntary, written consent to participate
* Current use of any pharmacotherapy for smoking cessation not provided by the researchers during the quit attempt
* Use of non-cigarette tobacco products as a primary form of tobacco use
* Being currently suicidal or homicidal
* Being medically unable to use the nicotine patch or nicotine gum/lozenge
* Psychotropic medication changes within 3 months of study initiation and during active treatment
* Current engagement in evidence-based therapies for PTSD or depression
* Pregnant or trying to become pregnant
* Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-09-08 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Cook, PhD, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (1):
- William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaye JT, Betts JM, Brubaker E, Webster K, Beckham JC, Baker TB, Cook JW. Behavioral Activation for Smoking Cessation in Veterans with Posttraumatic Stress Disorder: A Randomized Clinical Trial. Nicotine Tob Res. 2025 Aug 22;27(9):1524-1533. doi: 10.1093/ntr/ntaf054. PMID 40071390

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Behavioral Activation Therapy | Health and Smoking Education
Started | 63 | 61
Completed | 45 | 46
Not Completed | 18 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Activation Therapy | Health and Smoking Education | Total
Number analyzed (Participants) | 63 | 61 | 124
Age, Categorical [Count of Participants; unit: Participants] — Population: Missing age data from three participants.
  Participants
    number analyzed (Participants) | 61 | 60 | 121
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 55 | 54 | 109
    >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing age data from three participants.
  years
    number analyzed (Participants) | 61 | 60 | 121
    (all) | 50.70 (12.01) | 47.17 (13.02) | 48.95 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 52 | 57 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 61 | 59 | 120
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 7 | 11
  White | 54 | 52 | 106
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63 | 61 | 124
Baseline cigarettes smoked per day [Mean (Standard Deviation); unit: Cigarettes per day] | 18.67 (7.26) | 17.34 (8.26) | 17.99 (7.78)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Abstained From Smoking
Description: 7-day point prevalence abstinence at weeks 4, 12, 20, and 26 post target quit day
Time Frame: 26 weeks post target quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Activation Therapy | Health and Smoking Education
Number analyzed (Participants) | 63 | 61
Participants
  Week 4 | 23 | 21
  Week 12 | 20 | 19
  Week 20 | 22 | 14
  Week 26 | 12 | 8

2. Secondary Outcome: Time to Smoking Relapse
Description: Days to first relapse after the target quit date
Time Frame: 26 weeks post target quit date
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Behavioral Activation Therapy | Health and Smoking Education
Number analyzed (Participants) | 63 | 61
Days | 88.41 (73.46) | 84.34 (72.29)

3. Secondary Outcome: Clinician Administered PTSD Scale Score
Description: PTSD symptoms as assessed via the Clinician-Administered PTSD Scale (CAPS). Minimum score = 0, maximum score = 80. Higher scores indicate greater severity of symptoms.
Time Frame: 4 weeks post target quit date (end of treatment)
Population: Outcome Measure assessed at separate study visit. Data reported for participants who were assessed at this visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Behavioral Activation Therapy | Health and Smoking Education
Number analyzed (Participants) | 46 | 45
Units on a scale | 30.78 (11.80) | 27.33 (13.29)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 12 weeks post-target quit date while participants were taking study medication (nicotine patch and nicotine gum or lozenge).
Description: Study participants were asked: "Since our last contact, have there been any changes in your medical condition or health?" on the quit day, at weeks 1 through 4 post-quit, and at the 3-month follow up call. Participants also could self-initiate symptom reports during other phone calls.
Arm/Group | Behavioral Activation Therapy | Health and Smoking Education
All-Cause Mortality (participants affected / at risk) | 1/63 | 1/61
Serious Adverse Events (participants affected / at risk) | 7/63 | 6/61
Other Adverse Events (participants affected / at risk) | 33/63 | 29/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Activation Therapy (N=63) | Health and Smoking Education (N=61)
Hospitalized for chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalized for fall (General disorders) | 0 (0) | 1 (1)
Hospitalized for suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Hospitalized for shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Hospitalized for lightheadedness (Nervous system disorders) | 1 (1) | 0 (0)
Hospitalized for TIA (Nervous system disorders) | 0 (0) | 1 (1)
Hospitalized for wound care (Surgical and medical procedures) | 0 (0) | 1 (1)
Hospitalized for pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalized for back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Activation Therapy (N=63) | Health and Smoking Education (N=61)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 5 (7) | 8 (11)
Itching (Skin and subcutaneous tissue disorders) | 10 (10) | 11 (11)
Swelling or tingling of the mouth (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (3)
Skin rash (Skin and subcutaneous tissue disorders) | 7 (8) | 2 (4)
Insomnia (Psychiatric disorders) | 2 (2) | 5 (10)
Vivid dreams (Psychiatric disorders) | 10 (13) | 4 (10)
Hiccups (Gastrointestinal disorders) | 2 (2) | 2 (2)
Mouth problems (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1)
Persistent indigestion (Gastrointestinal disorders) | 8 (9) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT01995123/Prot_SAP_000.pdf